CLINICAL TRIAL: NCT01558206
Title: Bedside Ultrasonography of Chest Versus Pulmonary Artery CT Angiography in the Patients Who Came to Emergency Department of Alzahra General Hospital With Respiratory Symptoms and Signs in Favor of Pulmonary Thromboemboli.
Brief Title: Ultrasonography of Chest Versus Pulmonary Artery CT Angiography in Patients With Symptoms and Signs in Favor of PTE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Keihan Golshani, Assistant Professor of Emergency Medicine, Director of Emergency Medicine Residency Program, Isfahan University of Medical Sciences
Other Study IDs: 390327
Record Dates: First submitted 2012-03-08; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Thromboembolism
Keywords: PTE; Emergency bedside ultrasonography; pulmonary CT Angiography; Pulmonary Wedge infarction; Pulmonary Thromboembolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with impression of PTE: Those with signs and symptoms in favor of pulmonary thromboembolism.
  Interventions: Other: Pulmonary artery CT Angiography; Other: Emergency Bedside Ultrasonography of chest

INTERVENTIONS:
Other: Pulmonary artery CT Angiography — Performing Pulmonary artery CT Angiography for patients with signs and symptoms in favor of PTE.
Other: Emergency Bedside Ultrasonography of chest — Performing Emergency Bedside Ultrasonography of chest at the time of presentation for patients with signs and symptoms in favor of PTE.

SUMMARY:
In this study the investigators compare the diagnostic validity of Bedside Ultrasonography of chest and Pulmonary artery CT Angiography in the patients who came to Emergency Department of Alzahra General Hospital from 1 may 2012 to 1 October 2012 with respiratory symptoms and signs in favor of Pulmonary Thromboemboli (PTE).

ELIGIBILITY:
Inclusion Criteria:

* Patients with signs or symptoms in favor of PTE who come to Emergency department of Alzahra General Hospital.

Exclusion Criteria:

* previous history of Allergy to IV contrast
* Serum creatinin more than 1.8
* patients that will not agree to participate in the study.
* pregnancy
* Body weight more than 120 kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who come to the Emergency Department of Alzahra General Hospital with signs and symptoms in favor of PTE.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Emergency Ultrasonography findings in patients with signs and symptoms in favor of PTE. | Within 1 hour of admission
  Comparing the Emergency Bedside Ultrasonography findings in PTE with pulmonary CT Angiography findings.

SECONDARY OUTCOMES:
Pulmonary CT Angiography findings in patients with signs and symptoms in favor of PTE. | Within 24 hours of admission

CONTACTS AND LOCATIONS:
Overall Officials: Keihan Golshani, M.D., Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Emergency Department of alzahra General Hospital, Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran